CLINICAL TRIAL: NCT01978340
Title: Evaluation of EarlySense - a Contact-less Heart and Respiration Rate Monitor in Hospitalized Patients
Brief Title: Eval EarlySense Bet Lowenstein Sleeplab
Status: Withdrawn | Type: Observational
Sponsor: EarlySense Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: ES-CLC-2013_Prot_1
Record Dates: First submitted 2013-06-24; First posted 2013-11-07 (Estimated); Last update posted 2016-07-19 (Estimated); Status verified 2015-12

CONDITIONS: Obese; Sleep Apnea, Obstructive; Central Apnea; Sleep Disorders; Poor Quality Sleep
MeSH Terms: conditions — Obesity; Sleep Apnea, Obstructive; Sleep Apnea, Central; Sleep Wake Disorders

STUDY DESIGN:
Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: None Retained — no Biospeciments will be taken.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- sleeplab: Sleep Lab examined, usualy with some obesity or sleeping disorders.

SUMMARY:
The study objective is to collect heart rate, respiration rate and motion data of patients admitted to sleep lab and to determine the accuracy level of the EarlySense system vs. the monitors used in sleep lab (e.g., Polysomnography, respiratory belts, ECG, etc..) . Data regarding sleep condition, scoring and quality of sleep and in and out of bed status, patient turns will also be collected and compared to data collected by EarlySense contactless monitor. Different patient population will be monitored including obese, morbidly obese, patients with or without obstructive/central apnea, patients with or without arrhythmia as well as healthy population who arrive to sleep lab for general evaluation will be monitored

DETAILED DESCRIPTION:
EarlySense sensors will be placed under the mattress of subjects who have been included in the study. The sensors will not be in any contact with the patient. Two sensors will be utilized and placed under the subject's chest and pelvis area. Accuracy of the sensors will be compared to each other and to the reference device.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or above
2. Is willing to sign the consent form

Exclusion Criteria:

1. Age < 18 years
2. Is not willing to sign the consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Different patient population will be monitored including obese, morbidly obese, patients with or without apnea, patients with or without arrhythmia as well as healthy population who arrive to sleep lab for general evaluation will be monitored
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2013-11; Primary Completion 2014-02 (Estimated); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
To determine the accuracy level of the EarlySense system vs. the monitors used in sleep lab | up to 12 hours
  the measurements from the EarlySense System will be compared with the "Gold standard" equipment that is being used in the sleep Lab

CONTACTS AND LOCATIONS:
Overall Officials: Tatiana Vander, MD, Principal Investigator — Beit Lowenstein Hospital
Locations (1):
- Beit Lowenstien, Raa'nana, Israel